CLINICAL TRIAL: NCT04520828
Title: Immediate Effects of Postural Repositioning on Respiratory and Phonatory Tasks in Seated Individuals With Acquired Dysarthria: a Pilot Study
Brief Title: Immediate Effects of Postural Repositioning on Voice Production Tasks in Seated Individuals With Acquired Dysarthria:
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal (Other)
Responsible Party: Principal Investigator, Dorothy Barthélemy, Associate professor and researcher, Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROJET CRIR-722-0312
Record Dates: First submitted 2020-08-14; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Acquired Dysarthria (Finding)
Keywords: acquired dysarthria; corrected seated posture; maximum phonation duration; electromyographic patterns
MeSH Terms: conditions — Signs and Symptoms

STUDY DESIGN:
Intervention Model Description: pilot study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Postural repositioning (Experimental)
  Interventions: Other: postural repositioning

INTERVENTIONS:
Other: postural repositioning — The 10-min transdisciplinary intervention aimed (1) to facilitate and activate axial extension during standing and then during sitting; (2) to actively mobilize the trunk, cervical spine, and pelvic and shoulder girdles during standing and then during sitting; and (3) to adjust the seated position, as needed, with supports to ensure its maintenance throughout the experiment. Cushion, balls, boxes, or rolls were used to stabilize the final seated position.

SUMMARY:
To determine the effectiveness of a single 10-min postural repositioning session on the maximum phonation duration in individuals with acquired dysarthria.

DETAILED DESCRIPTION:
The impact of dysarthria goes beyond communication. However, there have been no clear directives guiding clinical practice to date, and despite increasing evidence directing treatment, research remains limited and predominantly consists of case studies or case series. Despite the importance of postural control in voice production, the effects of postural alignment on speech production efficiency are either little investigated or not at all explored in the dysarthric population. This study determined the effectiveness of a single 10-min postural repositioning session on the maximum phonation duration (MPD) in individuals with acquired dysarthria.

ELIGIBILITY:
**Participants with dysarthria Inclusion criteria

* sustained a stroke or traumatic brain injury
* diagnosed with dysarthria
* impaired postural control following a neurological injury
* are approaching the end of intensive rehabilitation or have finished intensive rehabilitation
* express a desire to participate in the research
* have the capacity to read.

Exclusion criteria

* had any cognitive impairment that could prevent them from understanding directives or from expressing their opinion about their posture A neurologist clinically assessed the cognitive function of PWDs

  **Control participants
* never diagnosed with dysarthria or any other voice impairment
* no comorbidities.
* no breathing deficits (e.g., asthma, chronic obstructive pulmonary disease)
* no pathologies in the spinal cord, spinal column, or thoracic cage that could prevent them from freely moving their trunk
* no neurological or cardiac problems.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-06-28 (Actual); Primary Completion 2015-07-16 (Actual); Study Completion 2015-07-16 (Actual)

PRIMARY OUTCOMES:
Change in maximum phonation duration | immediately before and after the 10 minute postural repositioning intervention
  Production of the vowel 'a' as long as possible without running out of air

SECONDARY OUTCOMES:
Change in trunk circumference in cm - Pre | immediately before postural repositioning intervention
  Measure of the circumference of the trunk taken at the level of the xyphoid process using a measuring tape when the participants achieves maximal inspiration and maximal expiration. The difference in circumference between maximal inspiration and maximal expiration is subsequently calculated.
Change in manometry | immediately before and after the 10 minute postural repositioning intervention
  time prolonged expiration
Change in EMG activation pattern | immediately before and after the 10 minute postural repositioning intervention
  pattern of electromyographic activity of muscles in the neck and trunk
Change in trunk circumference in cm - Post | immediately after the 10 minute postural repositioning intervention
  Measure of the circumference of the trunk taken at the level of the xyphoid process using a measuring tape when the participants achieves maximal inspiration and maximal expiration. The difference in circumference between maximal inspiration and maximal expiration is subsequently calculated.

OTHER OUTCOMES:
Change in the level of satisfaction of participants with their performance assessed using a questionnaire | immediately before and after the 10 minute postural repositioning intervention
  Following completion of voice tasks, the participants will be asked to grade their perceived level of performance in each posture (before and after the postural repositioning intervention) using the NER-21 scale. The participants are instructed to judge their vocal performance on the performance scale
Change in the participant's perceived effort to perform the task using a questionnaire | immediately before and after the 10 minute postural repositioning intervention
  Following completion of voice tasks, the participants will be asked to grade their effort in each posture (before and after the postural repositioning intervention) using the NER-21 scale. The participants are instructed to indicate the effort required to speak on the effort scale